CLINICAL TRIAL: NCT02258581
Title: A Long Term Follow-up Registry of Subjects Treated in A Gilead-Sponsored Trial in Subjects With Chronic Hepatitis B Infection
Brief Title: Long Term Follow-up Registry of Individuals Treated in A Gilead-Sponsored Trial in Individuals With Chronic Hepatitis B Infection
Status: Terminated | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-330-1508; 2015-001050-16 (EudraCT Number)
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — vesatolimod; Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GS-4774 — Exposure of interest for participants who received GS-4774 (administered as a subcutaneous injection) in a previous Gilead study for chronic hepatitis B virus infection.
Drug: GS-9620 — Exposure of interest for participants who received GS-9620 (tablets administered orally) in a previous Gilead study for chronic hepatitis B virus infection.
Drug: Tenofovir disoproxil fumarate (TDF) — Exposure of interest for participants who received TDF (tablets administered orally) in a previous Gilead study for chronic hepatitis B virus infection.
  Other Names: Viread®

SUMMARY:
This study will evaluate the long term effects of hepatitis B virus (HBV) treatment on the HBV serologic changes and HBV DNA levels through Week 144. This registry will enroll only individuals who were treated in a Gilead-sponsored trial for chronic hepatitis B (CHB).

ELIGIBILITY:
Key Inclusion Criteria:

* Must have participated in a Gilead-sponsored chronic hepatitis B (CHB) study no more than 120 days prior to Baseline (Day 1), except for participants from previous Gilead-sponsored study number GS-US-174-0149, who will have up to one year from their last visit in that protocol.
* Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Must be willing and able to comply with the visit schedule and study requirements
* Must have documented HBV DNA < 2,000 IU/mL at time of screening visit, which shall occur no later than 1 year post last study visit in GS-US-174-0149
* Must have documented hepatitis B surface antigen (HBsAg) negative status anytime during participation in GS-US-174-0149 regardless of ongoing HBV treatment

Key Exclusion Criteria:

* Patient participating or planning to participate in another clinical study with an investigational agent
* History of clinically-significant illness or any other major medical disorder that may interfere with follow-up, assessments or compliance with the protocol
* Believed by the Study Investigator to be inappropriate for study participation for any reason not otherwise listed
* Received TDF monotherapy either as part of GS-US-174-0149 Arm C (TDF monotherapy arm) or for TDF retreatment, and have taken any HBV antiviral therapy since completion of GS-US-174-0149

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who were treated in a Gilead-sponsored trial for hepatitis B virus infection.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with serum hepatitis B surface antigen (HBsAg) decline ≥ 0.5 log10 IU/ml from baseline at Week 48 | Week 48
  This endpoint will be measured for participants who are HBsAg positive at baseline.
Proportion of participants who remain HBsAg negative at Week 48 | Week 48
  This endpoint will be measured for participants who are HBsAg negative at baseline.

SECONDARY OUTCOMES:
Proportion of participants with serum HBsAg decline ≥ 0.5 log10 IU/ml from baseline at Week 144 | Week 144
  This endpoint will be measured for participants who are HBsAg positive at baseline.
Proportion of participants who achieve HBsAg loss at Weeks 48 and 144 | Weeks 48, 144
  This endpoint will be measured for participants who are HBsAg positive at baseline.
Proportion of participants who remain HBsAg negative at Week 144 | Week 144
  This endpoint will be measured for participants who are HBsAg negative at baseline.
Proportions of participants with hepatitis B envelope antigen (HBeAg) loss and seroconversion at Week 48 | Week 48
  This endpoint will be measured for participants who are HBeAg positive at baseline.
Proportions of participants with HBeAg loss and seroconversion at Week 144 | Week 144
  This endpoint will be measured for participants who are HBeAg positive at baseline.
Proportions of participants who remain HBeAg negative and hepatitis B envelope antibody (HBeAb) positive at Week 48 | Week 48
  This endpoint will be measured for HBeAg positive who achieved HBeAg seroconversion during the parental study.
Proportions of participants who remain HBeAg negative and HBeAb positive at Week 144 | Week 144
  This endpoint will be measured for HBeAg positive who achieved HBeAg seroconversion during the parental study.
Proportion of participants with HBV DNA < the lower limit of quantitation (LLOQ) at Weeks 48, 96 and 144 | Weeks 48, 96 and 144
  This endpoint will be measured for participants who are on treatment with oral antiviral (OAV) anti-HBV.
Change from Baseline in HBV DNA at Weeks 48, 96, and 144 | Baseline; Week 48; Week 96; Week 144

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (37):
- United States (16):
  - Kaiser Permanente, Sacramento, California
  - Kaiser Permanente, San Diego, California
  - Kaiser Permanente, San Francisco, California
  - Silicon Valley Research Institute, San Jose, California
  - University of Miami, Miami, Florida
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Digestive Disease Associates, PA, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. Louis University, St Louis, Missouri
  - Medical Procare, PLL, Flushing, New York
  - Northwell Health, Manhasset, New York
  - Xiaoli Ma, PC, Philadelphia, Pennsylvania
  - Bon Secours St. Mary's Hospital of Richmond, Newport News, Virginia
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Liver and Intestinal Research Centre, Vancouver, British Columbia
  - University of Manitoba, Winnepeg, Manitoba
  - Toronto General Hospital, Toronto, Ontario
- Hong Kong (2):
  - Princess Margaret Hospital, Lai Chi Kok
  - Prince of Wales Hospital, Shatin
- India (3):
  - Nirmal Hospital Private Limited, Surat, Gurarat
  - Midas Multispecialty Hospital Private Limited, Nagpur, Maharashtra
  - Dept. of Hepatology, School of Digestive & Liver Diseases, Kolkata, West Bengal
- Italy (4):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Universitaria Pisana, Caianello, Pisa
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria di Parma, Parma
- Auckland City Hospital, Auckland, New Zealand
- South Korea (5):
  - Pusan National, Busan
  - Korea University, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Yonsei University, Seoul